CLINICAL TRIAL: NCT00389025
Title: Mast-Cell Stabilizing Effects of Olopatadine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: C-05-30
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2010-01

CONDITIONS: Allergic Conjunctivitis
Keywords: Subject with clinical history of seasonal allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

INTERVENTIONS:
Drug: Olopatadine (generic name)

SUMMARY:
To assess the effects of olopatadine of the release of mast cell histamine

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic and not using any topical or systemic medication

Exclusion Criteria:

* Age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Tear histamine

SECONDARY OUTCOMES:
Tear cytology, subject evaluation of ocular itching, investigators evaluation of ocular redness

CONTACTS AND LOCATIONS:
Overall Officials: Terry Wiernas, Study Director — Alcon Research
Locations (1):
- Padova Site, Padua, Padova, Italy

REFERENCES:
- See also: Results on European Database — http://www.clinicaltrialsregister.eu/ctr-search/search?query=C-05-30